CLINICAL TRIAL: NCT03526029
Title: Observational Retrospective and Prospective Registry With Standardized Data Collection on Trauma Treatment in Switzerland
Brief Title: Swiss Trauma Registry
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-00331; ch18Jakob2
Record Dates: First submitted 2018-03-19; First posted 2018-05-16 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Trauma, Multiple; Trauma
MeSH Terms: conditions — Multiple Trauma; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Swiss Conference of Cantonal Health Directors has transferred the planning of highly specialized medicine to a specialized body under the direction of the Swiss Academy of Sciences. This specialist body has defined the treatment of critically ill as part of highly specialized medicine and founded the Swiss Trauma Registry at 12 hospitals in Switzerland. The registry is designed to provide a consistent and standardized approach and treatment outcomes in the short and long term quality control and as a basis for planning highly specialized medicine.

ELIGIBILITY:
Inclusion Criteria:

* injury severity code > 16 and 7 or abbreviated injury scale >3 for region of skull and brain

Exclusion Criteria:

* patients who will transferred in a burn unit
* drowned patients

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: severely injured patients at hospitals
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2040-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
mortality in severely injured patients | day of injury until year 5
  number of severely injured patients who died
patterns of injuries in severely injured patients | day of injury until year 5
  comparison of patterns of injuries in severely injured patients
Duration of primary hospitalisation after initial injury measured by days | day of injury until year 5
  Duration of primary hospitalisation after initial injury measured by days
Duration of secondary hospitalisation after initial injury measured by days | day of injury until year 5
  Duration of secondary hospitalisation after initial injury measured by days
Treatment costs in Swiss Francs | day of injury until year 5
  Treatment costs in Swiss Francs
line of treatments due to the initial injury (kind of treatment) | day of injury until year 5
  line of treatments due to the initial injury (kind of treatment)
line of treatments due to the initial injury (timepoints of treatments) | day of injury until year 5
  line of treatments due to the initial injury (timepoints of treatments)
Duration of Rehabilitation measured by days | day of injury until year 5
  Duration of Rehabilitation measured by days
Duration of incapacity for work measured by days | day of injury until year 5
  Duration of incapacity for work measured by days
diagnostic efforts measured by number and timepoint of imaging | day of injury until year 5
  number and timepoint of imaging
treatment efforts measured by number of medication given | day of injury until year 5
  number and timepoint of medication given and medical interventions performed
Primary supply Dates measured in minutes | on day of primary hospitalisation
  Primary supply Dates measured by time to start of surgery, time to admission to trauma room, time to ICU admission
treatment efforts measured by number of medical interventions performed | day of injury until year 5
  Treatment efforts measured by number and timepoint of medication given and medical interventions performed
treatment efforts measured by timepoint of medication given | day of injury until year 5
  Treatment efforts measured by number and timepoint of medication given and medical interventions performed
treatment efforts measured by timepoint of medical interventions performed | day of injury until year 5
  Treatment efforts measured by number and timepoint of medication given and medical interventions performed

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Marc Müller, Prof MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (12):
- Switzerland (12):
  - Kantonspital Aarau, Aarau
  - University Hospital Switzerland, Traumatology, Basel
  - Inselspital Bern, Bern
  - Kantonsspital Graubünden, Chur
  - University Hospital Geneva, Geneva
  - CHUV, Lausanne
  - Kantonsspital Luzern, Lucerne
  - Ospedale regionale die Lugano, Lugano
  - Kantonspital St.Gallen, Sankt Gallen
  - Gesundheitsnetz Wallis, Sion
  - Knatonsspital Winterthur, Winterthur
  - University Hospital Zürich, Zurich